CLINICAL TRIAL: NCT05382832
Title: Botox Vs Spinal Cord Stimulation in the Treatment of Refractory Migraine
Brief Title: Botox Vs Spinal Cord Stimulation in the Treatment of Refractory Migraine Clinical Trial
Acronym: BTX/SCS/TMig
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Europainclinics z.ú. (Other)
Collaborators: National Hospital for Neurology and Neurosurgery, London (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NSM 1-128/2021
Record Dates: First submitted 2022-05-04; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-Blinded, Randomized, Controlled Trial
Who Masked: Participant, Investigator
Masking Description: In order to have a double-blinded RCT, the investigators will not be aware of the trial branch of the participants. Injections will be performed either with Botulinum Toxin or with Normal Saline and Spinal Cord Stimulators will be configured in order to use high-frequency stimulation or a sham treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A1 Group SCS (Experimental): Botox Injection and the SCS Internal Pulse Generator turned on in sham-mode. Starting two weeks after the SCS implant
  Interventions: Combination Product: SCS
- A1 Group Botox (Experimental): Botox Injection and the SCS Internal Pulse Generator turned on in sham-mode. Starting two weeks after the SCS implant
  Interventions: Combination Product: SCS
- B1 Group SCS (Placebo Comparator): Placebo Injection and Internal Pulse Generator turned on in the high-frequency working mode. Starting two weeks after the SCS implant
  Interventions: Combination Product: SCS
- B1 Group Saline (Placebo Comparator): Placebo Injection and Internal Pulse Generator turned on in the high-frequency working mode. Starting two weeks after the SCS implant
  Interventions: Combination Product: SCS
- A2 Group SCS (Experimental): Botox Injection and the SCS Internal Pulse Generator turned on in sham-mode. Starting at the 28th week of clinical trial investigation
  Interventions: Combination Product: SCS
- A2 Group Botox -after washout period (Experimental): Botox Injection and the SCS Internal Pulse Generator turned on in sham-mode. Starting at the 28th week of clinical trial investigation
  Interventions: Combination Product: SCS
- B2 Group SCS (Placebo Comparator): Placebo Injection and Internal Pulse Generator turned on in the high-frequency working mode. Starting at the 28th week of clinical trial investigation
  Interventions: Combination Product: SCS
- B2 Group Saline -after washout period (Placebo Comparator): Placebo Injection and Internal Pulse Generator turned on in the high-frequency working mode. Starting at the 28th week of clinical trial investigation
  Interventions: Combination Product: SCS

INTERVENTIONS:
Combination Product: SCS — SCS-experimental treatment
  Other Names: Botox
Combination Product: SCS — SCS-placebo
  Other Names: Saline

SUMMARY:
The clinical trial is focused on the treatment of selected patients with a migraine after implantation of spinal cord stimulator (SCS) based on previous neurological examination. Patients will be randomized and divided into two groups. According to randomization patients will receive saline or botox into the epidural space. The efficacy of treatment will be compared and estimated in both groups during different SCS settings. Data will be collected in pre-set time frames.

DETAILED DESCRIPTION:
This study consists of a double-blind randomized cross-over controlled trial (RCT). Enrolled centers are National Hospital For Neurology and Neurosurgery in London in the United Kingdom, EuroPainClinics® with centers in Bratislava, Košice, and Bardejov in the Slovac republic and also EuroPainClinics® with centers Praha, Brno, Ostrava, and Hradec Kralove in the Czech republic.

Patients with diagnosing migraine (examined previously by neurologist) suitable for participating in the clinical trial, without any previous Botulinum Toxin treatment or Spinal Cord Stimulation therapy, (after exact consultation by neuromodulation team) will be offered to enroll in the BoStiM trial.

Enrolled patients will have a full implant of Nevro Senza SCS system. The intervention will be performed at the National Hospital for Neurology and Neurosurgery in London in the United Kingdom, and also in st. Michal Hospital in Bratislava in the Slovak Republic and General University Hospital in Prague in the Czech Republic. The procedure will be performed by the Neuromodulation Team. The implanted SCS will be turned off at this stage and will stay off for 2 weeks' time to let the wounds heal properly and not interfere with headache measurements. Once enrolled in the study, the patients will be randomized into one of the two groups of study. Groups will consist in either first SCS treatment, then washout period, then Botox treatment or SCS, then washout, then Botox. All patients will therefore be their own controls, and all of them will receive both treatments. After randomization, patients will be added to the SCS pathway. During the period between enrolment and SCS implant, patients will have the opportunity to meet the psychology team at the Pain Management Centre (PMC) and will undergo teaching sessions to learn the basic SCS practical aspects.

Blinding technique:

In order to have a double-blinded RCT, the investigators will not be aware of the trial branch of the participants.

Injections will be performed either with Botulinum Toxin or with Normal Saline and Spinal Cord Stimulators will be configured in order to use high-frequency stimulation or a sham treatment. All Internal Pulse Generators (IPG) will be turned on throughout the trial so as to avoid the participants being able to know the treatment they're really receiving at that time. Participants receiving Botox injections will have their IPG running with a sham configuration. They will not be receiving any electric stimulation over the leads, but the battery will be programmed to have a current leakage and will need to be recharged so as if the IPG was properly working. This again is to avoid them knowing which treatment they're receiving at any time being. The Clinical Specialist Nurses (CNS) of our PMC will be in charge of labeling the Botox/Placebo vials, which will be anonymized, and they will also be in charge of setting up the SCS (sham or treatment).

Data collection:

The enrolled patients will be provided a Smartphone to assess the migraine episodes. Each Smartphone will have an in-built app that the patients will use daily, and that will send the results to the research team. Those patients preferring to use their own smartphone will need to download the app to their smartphone. The app will include a visual numeric scale (VNS) that the participants will need to fulfill daily, as well as qualitative questions including the type of migraine, the onset, presence or absence of aura, duration of the episode, and possible medication intake.

The first period of trial:

The proper trial period will start two weeks after the implant (week 1). On this day, patients will be invited to come to the PMC. Depending on the randomization group, patients will have either a Botox Injection and the SCS Internal Pulse Generator turned on in sham-mode or a placebo injection and the IPG turned on in proper working mode. Patients will be given a controller for the IPG so that they may be able to turn it off in case of an emergency. They will nonetheless not be able to change the program. None of the investigators will be aware of the group. At week 12, participants will have a new injection of either Botox or Placebo and will be reviewed by the CNS and Nevro team to assess any problems. At that time, they will also be asked to complete through the Smartphone app the Quality of Life (QoL) questionnaires and will be asked to guess their branch. Washout period: At week 24, all participants will undergo a washout period of 1 month. They will be invited to come to the PMC and IPG (both sham and treatment) will be turned off. They will also be asked to fill the QoL questionnaires.

Second Period of Trial:

At week 28, participants will be invited to come to the PMC and they will start the second part of the trial, being assigned to the other branch. All IPG's will be turned on, those previously being actively treating will be turned to the sham mode and the opposite will be done with previously sham mode ones. Patients previously receiving placebo injections will receive a Botox injection on that day, and those previously receiving Botox injections will receive a placebo one. Quality of life questionnaires will be filled. At week 40, participants will undergo the 4th and last series of injections (Botox or placebo) and will have an assessment with CNS and Nevro team, and will be asked to fill in the usual questionnaires.

End of trial:

The trial will end at week 52 when patients will be asked to fill in the usual questionnaires. At that moment, they will be communicated to which branch they had been assigned.

Patients will then decide whether they want to keep the SCS system or prefer it removed.

ELIGIBILITY:
Inclusion Criteria:

* migraine presence

Exclusion Criteria:

* disagreement with participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Health Questionnaire (EQ-5D-5L) | 14 days after the SCS implant
  1 Graded from 1-5, where 1 means no problems in the area and 5 meaning extreme problems
Health Questionnaire (EQ-5D-5L) | 91 days after the SCS implant
  Week 13 Graded from 1-5, where 1 means no problems in the area and 5 meaning extreme problems
Health Questionnaire (EQ-5D-5L) | 175 days after the SCS implant
  Week 25 Graded from 1-5, where 1 means no problems in the area and 5 meaning extreme problems
Health Questionnaire (EQ-5D-5L) | 196 days after the SCS implant
  Week 28 Graded from 1-5, where 1 means no problems in the area and 5 meaning extreme problems
Health Questionnaire (EQ-5D-5L) | 280 days after the SCS implant
  Week 40 Graded from 1-5, where 1 means no problems in the area and 5 meaning extreme problems
Health Questionnaire (EQ-5D-5L) | 364 dayss after the SCS implant
  Week 52

SECONDARY OUTCOMES:
Visual numeric scale | daily up to 10 days
Type of migraine | up to 1 week
Aura presence | up to 1 week
Duration of the migraine episode | up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Róbert Rapcan, MD, PhD, MBA, FIPP, Study Chair — EuroPainClincs; Ladislav Kočan, MD, PhD, Study Chair — EuroPainClincs